CLINICAL TRIAL: NCT06552689
Title: First Human Study of Sutra Hemi-Valve to Evaluate Safety and Efficacy in Patients With Mitral Regurgitation
Brief Title: Sutra Hemi-valve First-in-Human Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sutra Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-002
Record Dates: First submitted 2024-08-06; First posted 2024-08-14 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Mitral Regurgitation
Keywords: mitral regurgitation; transcatheter mitral valve replacement; transcatheter mitral valve repair; hemi-valve
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sutra Hemi-valve Transcatheter Mitral Valve Replacement (TMVR) (Experimental): The Sutra Hemi-valve TMVR System is an innovative approach developed as a treatment for mitral regurgitation consisting of the Sutra Hemi-valve posterior leaflet replacement device, and the 32 Fr trans-septal delivery system.
  Interventions: Device: Sutra Hemi-valve Transcatheter Mitral Valve Replacement (TMVR) System

INTERVENTIONS:
Device: Sutra Hemi-valve Transcatheter Mitral Valve Replacement (TMVR) System — Trans-septal Sutra Hemi-valve TMVR System to treat mitral regurgitation

SUMMARY:
Study to evaluate the feasibility, safety and performance of the Sutra Hemi-valve Transcatheter Mitral Valve Replacement System in patients with moderate-severe and severe symptomatic mitral regurgitation who are at high risk for surgical treatment.

DETAILED DESCRIPTION:
Investigational Device:

Sutra Transcatheter Mitral Valve Replacement (TMVR) System The Sutra Hemi-valve TMVR System consists of 32Fr delivery devices and an implantable hemi-valve.

The Sutra Hemi-valve consists of a self-expanding nitinol frame, a tri-leaflet bovine pericardial hemi-valve, and a sealing skirt. The Sutra Hemi-valve is intended to replace the posterior leaflet of the mitral valve to treat mitral regurgitation. The frame consists of an atrial portion for anchoring to the native annulus, and a ventricular portion which houses the Hemi-valve. The atrial section of the Sutra Hemi-valve contains three through-holes for anchoring to Dual-guiding-and-fixation (DGF) devices implanted at the lateral trigone (T1), the medial trigone (T3), and in the center of the posterior annulus (P2). The Sutra Hemi-valve comes in two sizes: Size 42 and Size 38.

Intended Use: The Sutra Hemi-valve TMVR system is intended for use as a partial replacement mitral valve.

Indication for Use: The Sutra Hemi-valve TMVR system is indicated for use in patients with moderate-severe or severe symptomatic mitral regurgitation who are considered high risk for conventional mitral valve surgery.

Trial Design: Prospective, multi-center, unblinded, single arm first in human/ feasibility clinical study.

Primary Objective:

To assess the safety and performance of the Sutra Hemi-valve TMVR System in patients with moderate-severe or severe symptomatic mitral regurgitation who are considered high risk for conventional mitral valve surgery.

Secondary Objectives:

* Improvement of mitral regurgitation
* Assess interaction of implant prosthesis with native mitral valve apparatus, conduction system, left ventricular outflow tract (LVOT) and aortic valve
* Assess stability of implant.
* Assess hemodynamics of the mitral valve apparatus

ELIGIBILITY:
Inclusion Criteria:

* Subject is greater than 18 years of age at time of enrollment.
* Subject has moderate-severe or severe symptomatic mitral regurgitation who are considered high surgical risk for conventional mitral repair or replacement, as assessed by institutional multidisciplinary heart team.
* New York Heart Association (NYHA) Functional Class II and above.
* Subject anatomy is suitable for transfemoral and transeptal device delivery and meets sizing criteria for Sutra Hemi-valve TMVR System.
* Subject willing and able to provide informed consent and able to comply with the study protocol and follow up.
* Female subjects of childbearing potential have a negative pregnancy test ≤ 7 days before the procedure

Exclusion Criteria:

* Prohibitive mitral annular calcification
* Diseased mitral anterior leaflet such as flail or prolapse
* Previous mitral valve intervention
* Implanted with venous stents (iliac and femoral) including inferior vena cava (IVC) filter or congenital abnormalities of the IVC that would preclude ability for transfemoral access with the delivery system.
* Evidence of intra-cardiac, inferior vena cava (IVC) or ipsilateral femoral venous thrombus
* Severe aortic stenosis or insufficiency (Note: may be treated ≥ 30 days prior to study procedure)
* Contraindication for transesophageal echocardiography (TEE) or MDCT scan
* Active infections requiring current antibiotic therapy (if temporary illness, patients may enroll 2 weeks after discontinuation of antibiotics)
* Endocarditis within 6 months
* Left ventricular ejection fraction (LVEF) < 25%
* Severe Chronic Obstructive Pulmonary Disease (COPD) demonstrated by Forced Expiratory Volume (FEV1) < 750cc
* Implant or revision of any pacing device < 30 days prior to intervention
* Symptomatic coronary artery disease treated < 30 days prior to study procedure
* Active peptic ulcer or upper gastrointestinal bleeding within 90 days
* Prior stroke, TIA, or myocardial infarction within 90 days
* Severe renal insufficiency (creatinine > 225 µmol/L) or patient requiring dialysis
* Any endovascular therapeutic interventional or surgical procedure performed within 30 days prior to enrollment
* Pregnant, nursing or planning to be pregnant. (Female participants of childbearing potential must have a negative pregnancy test prior to enrollment)
* History of bleeding diathesis or coagulopathy that cannot be managed or patient will refuse blood transfusion
* Hemodynamic instability requiring dependency on either inotropic agents or mechanical circulatory support
* Known hypersensitivity or contraindication to heparin and bivalirudin
* Known allergy to nitinol or contrast agents that cannot be pre-medicated
* Severe dementia or lack of capacity due to conditions that result in either inability to provide informed consent for the trial/procedure, prevent independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up assessments.
* Patient is participating in another investigational drug or device clinical study that has not completed primary endpoint follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint - The ability of the Sutra Hemi-valve to be placed without Major Device Related Adverse Events through thirty (30) days | Day 30
  including:
  * Death (Cardiovascular mortality vs non-cardiovascular);
  * Reintervention (operative or transcatheter) due to progressive or recurrent MR or device related complications;
  * Disabling stroke;
  * Myocardial infarction (MVARC);
  * Major access site and vascular complications;
  * Fatal or life-threatening bleeding (MVARC Type III-V);
  * Renal Failure requiring dialysis;
  * Cardiac tamponade.
Primary Performance Endpoint - Sutra Hemi-valve TMVR System Technical Success | Day 0
  defined as: successful access, delivery, and retrieval of the delivery system; and successful deployment and correct positioning of the implant; and no need for additional emergency surgery or re-intervention related to the investigational device or index procedure.

SECONDARY OUTCOMES:
Intra-procedure MR severity is reduced by at least 1 grade from baseline per echo (e.g., from severe to moderate). | Day 0
Post-index procedure (discharge or within 7 Days post-index procedure, whichever is earliest) MR severity is reduced by at least 1 grade from baseline per echo (e.g., from severe to moderate). | Day 0 - Day 7
MR severity grade per Echo | Day 30, Month 6, Month 12
Change in NYHA functional class | Day 30, Month 6, Month 12
6 Minute Walk Test distance (6MWT) | Day 30, Month 6, Month 12

OTHER OUTCOMES:
Change in LV ejection fraction | Day 30, Month 6, Month 12
Change in LV end diastolic volume index (LVEDVI) | Day 30, Month 6, Month 12
Change in LV end systolic volume index (LVESVI) | Day 30, Month 6, Month 12
Change in LV stroke volume | Day 30, Month 6, Month 12
Heart failure hospitalizations | Day 30, Month 6, Month 12
Number of days alive and out of hospital | Day 30, Month 6, Month 12

CONTACTS AND LOCATIONS:
Locations (1):
- Waikato Hospital, Hamilton, New Zealand

IPD SHARING:
Plan to Share IPD: No